CLINICAL TRIAL: NCT02422511
Title: Genomic Sequencing for Childhood Risk and Newborn Illness (The BabySeq Project)
Brief Title: Genomic Sequencing for Childhood Risk and Newborn Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Boston Children's Hospital (Other); Baylor College of Medicine (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Human Genome Research Institute (NHGRI) (NIH); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Robert C. Green, MD, MPH, Professor of Medicine, Division of Genetics, Department of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: The BabySeq Project; U19HD077671 (NIH)
Record Dates: First submitted 2015-04-10; First posted 2015-04-21 (Estimated); Results first posted 2021-08-31 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Hereditary Disease; Genetic Predisposition to Disease
Keywords: Genome Sequencing; Exome Sequencing; Newborn Screening; Childhood Onset Genetic Conditions
MeSH Terms: conditions — Genetic Diseases, Inborn; Genetic Predisposition to Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: Families are masked to randomization until disclosure sessions
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Well Baby Family History Only (Active Comparator): Parents of newborns in well-baby units receive an Annotated Family History Report only. Active Comparator: Standard of Care Only: Family History report only
  Interventions: Other: Family history report
- Well Baby Family History + Exome Sequencing (Experimental): Parents of newborns in well-baby units receive a Genome Report and an Annotated Family History Report. Main Study Experimental: Genome Report and Family History report
  Interventions: Genetic: Genomic sequencing; Other: Family history report
- ICU Baby Family History Only (Active Comparator): Parents of newborns in intensive care units receive an Annotated Family History Report only. Active Comparator: Standard of Care Only: Family History report only
  Interventions: Other: Family history report
- ICU Baby Family History + Exome Sequencing (Experimental): Parents of newborns in intensive care units receive a Genome Report and an Annotated Family History Report. Main Study Experimental: Genome Report and Family History report
  Interventions: Genetic: Genomic sequencing; Other: Family history report

INTERVENTIONS:
Genetic: Genomic sequencing — Both sick and healthy infants randomized to receive genomic sequencing will receive a 'Genomic Newborn Sequencing Report' (GNSR) which will include pathogenic or likely pathogenic variants identified in genes associated with childhood-onset disease.
  Arms: ICU Baby Family History + Exome Sequencing; Well Baby Family History + Exome Sequencing
Other: Family history report — Participants from all arms of the study will have a family history taken by a study genetic counselor. Information collected through the family history will be summarized in a family history report that will be reviewed with all participants.

SUMMARY:
The Genomic Sequencing for Childhood Risk and Newborn Illness (the BabySeq Project) is a research study exploring the use of genomic sequencing in newborns. The National Institutes of Health is funding this study.

The investigators will enroll 240 healthy infants and their parents from the Brigham and Women's Hospital (BWH) Well Newborn Nursery and 240 sick infants and their parents at Boston Children's Hospital (BCH) or the BWH Neonatal Intensive Care Unit (NICU). A small blood sample will be collected from each infant and genome sequencing may be performed. Six weeks later, results are returned and explained. Over 12 months the investigators are studying the experiences of parents and pediatricians of infants who receive sequencing to help understand how best to use genomics in pediatric care.

DETAILED DESCRIPTION:
The objective of this research protocol is to conduct a randomized clinical trial to assess the benefits and risks of adding the information from a genomic sequencing report to physician-mediated medical care of newborns during their pediatric years.

The investigators will enroll 240 healthy infants and their parents from the Brigham and Women's Hospital (BWH) Well Newborn Nursery and 240 sick infants and their parents at Boston Children's Hospital (BCH) or the BWH Neonatal Intensive Care Unit (NICU).

A small blood sample will be obtained from each enrolled infant. Samples will be collected from all infants enrolled, regardless of the arm to which they are assigned, in order to follow the same protocol for all subjects prior to randomization.

Infants within each cohort will be randomized (1:1) to either standard-of-care (family history and standard newborn screening report) or to standard-of-care plus genomic sequencing.

A study physician and genetic counselor will disclose the infant's randomization assignment and study results during an in-person consultation with each family. The study physician and genetic counselor will provide the consultation to families utilizing all available medical information. In the sequencing arm of the study, this will include the medical history, physical exam, family history, standard newborn screening (NBS) report and sequencing report(s). In the non-sequencing arm of the study, this will include the medical history, physical exam, family history and standard NBS report.

Parents will be surveyed at four points over the 12 months after enrollment: baseline, immediately post-disclosure (approximately 6 weeks after enrollment), 3 months post-disclosure, and at 10 months post-disclosure.

ELIGIBILITY:
Newborns and Parents at Brigham and Women's Hospital (BWH) Well Newborn Nursery:

Inclusion Criteria :

1. Infants born at BWH and admitted to the Well Newborn Nursery
2. At least one biological parent is physically available to have genetic counseling, donate DNA, and provide consent for testing the infant. If the second biological parent is known but not physically present, the second biological parent must be available to have genetic counseling by phone, return a signed consent form by mail, and donate DNA via a mailed saliva kit. If there is a "rearing parent" (an individual who is not biologically related to the infant, but who is dedicated to raising the child), that individual must also provide consent but will not be asked to submit a saliva sample.
3. Mother (either rearing or biological) carried the pregnancy

Exclusion Criteria:

1. Parents are non-English speaking
2. Parents are unwilling to have genomic reports placed in the medical record or sent to their primary care pediatrician
3. Mother or father younger than 18 years of age
4. Mother or father with impaired decisional capacity
5. Age of infant is older than 30 days
6. One of a multiple gestation
7. Any infant in which clinical considerations preclude drawing 1.0 ml of blood
8. Missing consent of either biological parent (if known) or rearing parent (if applicable)

Sick Newborns and Parents at Boston Children's Hospital (BCH) or the BWH NICU:

Inclusion Criteria:

1. Infants admitted to BCH or the BWH NICU
2. At least one biological parent is physically available to have genetic counseling, donate DNA, and provide consent for testing the infant. If the second biological parent is known but not physically present, the second biological parent must be available to have genetic counseling by phone, return a signed consent form by mail, and donate DNA via a mailed saliva kit. If there is a "rearing parent" (an individual who is not biologically related to the infant, but who is dedicated to raising the child), that individual must also provide consent but will not be asked to submit a saliva sample.
3. Mother (either biological or rearing) carried the pregnancy

Exclusion Criteria:

1. Parents are non-English speaking
2. Parents are unwilling to have genomic reports placed in the medical record or sent to their primary care pediatrician
3. Mother or father younger than 18 years of age
4. Mother or father with impaired decisional capacity
5. Age of infant is older than 30 days
6. One of a multiple gestation
7. Any infant in which clinical considerations preclude drawing 1.0 ml of blood
8. Hospital admission expected to be less than 72 hours
9. Missing consent of either biological parent (if known) or rearing parent (if applicable)
10. Previously performed exome/genome sequencing on patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1205 (Actual)
Dates: Start 2015-05; Primary Completion 2020-04 (Actual); Study Completion 2021-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Green, MD, MPH, Principal Investigator — Brigham and Women's Hospital; Alan Beggs, PhD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

REFERENCES:
- [Background] Waisbren SE, Back DK, Liu C, Kalia SS, Ringer SA, Holm IA, Green RC. Parents are interested in newborn genomic testing during the early postpartum period. Genet Med. 2015 Jun;17(6):501-4. doi: 10.1038/gim.2014.139. Epub 2014 Dec 4. PMID 25474344
- [Background] Green RC, Rehm HL, Kohane IS. Clinical genome sequencing. In: Ginsburg GS, Willard HF, eds. Genomic and Personalized Medicine. Vol 1. 2nd ed. San Diego: Academic Press; 2013: 102-122.
- [Background] Dewey FE, Grove ME, Pan C, Goldstein BA, Bernstein JA, Chaib H, Merker JD, Goldfeder RL, Enns GM, David SP, Pakdaman N, Ormond KE, Caleshu C, Kingham K, Klein TE, Whirl-Carrillo M, Sakamoto K, Wheeler MT, Butte AJ, Ford JM, Boxer L, Ioannidis JP, Yeung AC, Altman RB, Assimes TL, Snyder M, Ashley EA, Quertermous T. Clinical interpretation and implications of whole-genome sequencing. JAMA. 2014 Mar 12;311(10):1035-45. doi: 10.1001/jama.2014.1717. PMID 24618965
- [Background] Gilissen C, Hoischen A, Brunner HG, Veltman JA. Unlocking Mendelian disease using exome sequencing. Genome Biol. 2011 Sep 14;12(9):228. doi: 10.1186/gb-2011-12-9-228. PMID 21920049
- [Background] Gonzaga-Jauregui C, Lupski JR, Gibbs RA. Human genome sequencing in health and disease. Annu Rev Med. 2012;63:35-61. doi: 10.1146/annurev-med-051010-162644. PMID 22248320
- [Background] The President's Council on Bioethics. The changing moral focus of newborn screening: An ethical analysis by the President's Council on Bioethics. 2008; http://bioethics.georgetown.edu/pcbe/reports/newborn_screening.
- [Background] Saunders CJ, Miller NA, Soden SE, Dinwiddie DL, Noll A, Alnadi NA, Andraws N, Patterson ML, Krivohlavek LA, Fellis J, Humphray S, Saffrey P, Kingsbury Z, Weir JC, Betley J, Grocock RJ, Margulies EH, Farrow EG, Artman M, Safina NP, Petrikin JE, Hall KP, Kingsmore SF. Rapid whole-genome sequencing for genetic disease diagnosis in neonatal intensive care units. Sci Transl Med. 2012 Oct 3;4(154):154ra135. doi: 10.1126/scitranslmed.3004041. PMID 23035047
- [Background] Yang Y, Muzny DM, Reid JG, Bainbridge MN, Willis A, Ward PA, Braxton A, Beuten J, Xia F, Niu Z, Hardison M, Person R, Bekheirnia MR, Leduc MS, Kirby A, Pham P, Scull J, Wang M, Ding Y, Plon SE, Lupski JR, Beaudet AL, Gibbs RA, Eng CM. Clinical whole-exome sequencing for the diagnosis of mendelian disorders. N Engl J Med. 2013 Oct 17;369(16):1502-11. doi: 10.1056/NEJMoa1306555. Epub 2013 Oct 2. PMID 24088041
- [Background] Biesecker LG, Green RC. Diagnostic clinical genome and exome sequencing. N Engl J Med. 2014 Sep 18;371(12):1170. doi: 10.1056/NEJMc1408914. No abstract available. PMID 25229935
- [Background] Vassy JL, Lautenbach DM, McLaughlin HM, Kong SW, Christensen KD, Krier J, Kohane IS, Feuerman LZ, Blumenthal-Barby J, Roberts JS, Lehmann LS, Ho CY, Ubel PA, MacRae CA, Seidman CE, Murray MF, McGuire AL, Rehm HL, Green RC; MedSeq Project. The MedSeq Project: a randomized trial of integrating whole genome sequencing into clinical medicine. Trials. 2014 Mar 20;15:85. doi: 10.1186/1745-6215-15-85. PMID 24645908
- [Background] Holm IA, Savage SK, Green RC, Juengst E, McGuire A, Kornetsky S, Brewster SJ, Joffe S, Taylor P. Guidelines for return of research results from pediatric genomic studies: deliberations of the Boston Children's Hospital Gene Partnership Informed Cohort Oversight Board. Genet Med. 2014 Jul;16(7):547-52. doi: 10.1038/gim.2013.190. Epub 2014 Jan 9. PMID 24406460
- [Background] Comeau AM, Parad RB, Dorkin HL, Dovey M, Gerstle R, Haver K, Lapey A, O'Sullivan BP, Waltz DA, Zwerdling RG, Eaton RB. Population-based newborn screening for genetic disorders when multiple mutation DNA testing is incorporated: a cystic fibrosis newborn screening model demonstrating increased sensitivity but more carrier detections. Pediatrics. 2004 Jun;113(6):1573-81. doi: 10.1542/peds.113.6.1573. PMID 15173476
- [Background] Wilfond BS, Parad RB, Fost N. Balancing benefits and risks for cystic fibrosis newborn screening: implications for policy decisions. J Pediatr. 2005 Sep;147(3 Suppl):S109-13. doi: 10.1016/j.jpeds.2005.08.019. PMID 16202773
- [Background] Bhattacharjee A, Sokolsky T, Wyman SK, Reese MG, Puffenberger E, Strauss K, Morton H, Parad RB, Naylor EW. Development of DNA confirmatory and high-risk diagnostic testing for newborns using targeted next-generation DNA sequencing. Genet Med. 2015 May;17(5):337-47. doi: 10.1038/gim.2014.117. Epub 2014 Sep 25. PMID 25255367
- [Background] Connolly M, Holm I, Beggs A, Agrawal P. Bringing current research technology to the clinic: The Manton Center for Orphan Disease Research Gene Discovery Core (Platform Abstract/Program 45). Paper presented at: 12th International Congress of Human Genetics/61st Annual Meeting of The American Society of Human Genetics; October 12, 2011, 2011; Montreal, Canada.
- [Background] McGuire AL, Caulfield T, Cho MK. Research ethics and the challenge of whole-genome sequencing. Nat Rev Genet. 2008 Feb;9(2):152-6. doi: 10.1038/nrg2302. PMID 18087293
- [Background] Waisbren SE, Levy HL. Expanded screening of newborns for genetic disorders. JAMA. 2004 Feb 18;291(7):820-1; author reply 821. doi: 10.1001/jama.291.7.820-c. No abstract available. PMID 14970058
- [Background] Berg JS, Agrawal PB, Bailey DB Jr, Beggs AH, Brenner SE, Brower AM, Cakici JA, Ceyhan-Birsoy O, Chan K, Chen F, Currier RJ, Dukhovny D, Green RC, Harris-Wai J, Holm IA, Iglesias B, Joseph G, Kingsmore SF, Koenig BA, Kwok PY, Lantos J, Leeder SJ, Lewis MA, McGuire AL, Milko LV, Mooney SD, Parad RB, Pereira S, Petrikin J, Powell BC, Powell CM, Puck JM, Rehm HL, Risch N, Roche M, Shieh JT, Veeraraghavan N, Watson MS, Willig L, Yu TW, Urv T, Wise AL. Newborn Sequencing in Genomic Medicine and Public Health. Pediatrics. 2017 Feb;139(2):e20162252. doi: 10.1542/peds.2016-2252. Epub 2017 Jan 17. PMID 28096516
- [Background] Ceyhan-Birsoy O, Machini K, Lebo MS, Yu TW, Agrawal PB, Parad RB, Holm IA, McGuire A, Green RC, Beggs AH, Rehm HL. A curated gene list for reporting results of newborn genomic sequencing. Genet Med. 2017 Jul;19(7):809-818. doi: 10.1038/gim.2016.193. Epub 2017 Jan 12. PMID 28079900
- [Background] Murry JB, Machini K, Ceyhan-Birsoy O, Kritzer A, Krier JB, Lebo MS, Fayer S, Genetti CA, VanNoy GE, Yu TW, Agrawal PB, Parad RB, Holm IA, McGuire AL, Green RC, Beggs AH, Rehm HL; BabySeq Project Team. Reconciling newborn screening and a novel splice variant in BTD associated with partial biotinidase deficiency: a BabySeq Project case report. Cold Spring Harb Mol Case Stud. 2018 Aug 1;4(4):a002873. doi: 10.1101/mcs.a002873. Print 2018 Aug. PMID 29728376
- [Background] Holm IA, Agrawal PB, Ceyhan-Birsoy O, Christensen KD, Fayer S, Frankel LA, Genetti CA, Krier JB, LaMay RC, Levy HL, McGuire AL, Parad RB, Park PJ, Pereira S, Rehm HL, Schwartz TS, Waisbren SE, Yu TW; BabySeq Project Team; Green RC, Beggs AH. The BabySeq project: implementing genomic sequencing in newborns. BMC Pediatr. 2018 Jul 9;18(1):225. doi: 10.1186/s12887-018-1200-1. PMID 29986673
- [Background] Genetti CA, Schwartz TS, Robinson JO, VanNoy GE, Petersen D, Pereira S, Fayer S, Peoples HA, Agrawal PB, Betting WN, Holm IA, McGuire AL, Waisbren SE, Yu TW, Green RC, Beggs AH, Parad RB; BabySeq Project Team. Parental interest in genomic sequencing of newborns: enrollment experience from the BabySeq Project. Genet Med. 2019 Mar;21(3):622-630. doi: 10.1038/s41436-018-0105-6. Epub 2018 Sep 13. PMID 30209271
- [Background] Ceyhan-Birsoy O, Murry JB, Machini K, Lebo MS, Yu TW, Fayer S, Genetti CA, Schwartz TS, Agrawal PB, Parad RB, Holm IA, McGuire AL, Green RC, Rehm HL, Beggs AH; BabySeq Project Team. Interpretation of Genomic Sequencing Results in Healthy and Ill Newborns: Results from the BabySeq Project. Am J Hum Genet. 2019 Jan 3;104(1):76-93. doi: 10.1016/j.ajhg.2018.11.016. PMID 30609409
- [Background] Pereira S, Robinson JO, Gutierrez AM, Petersen DK, Hsu RL, Lee CH, Schwartz TS, Holm IA, Beggs AH, Green RC, McGuire AL; BabySeq Project Group. Perceived Benefits, Risks, and Utility of Newborn Genomic Sequencing in the BabySeq Project. Pediatrics. 2019 Jan;143(Suppl 1):S6-S13. doi: 10.1542/peds.2018-1099C. PMID 30600265
- [Background] Holm IA, McGuire A, Pereira S, Rehm H, Green RC, Beggs AH; BabySeq Project Team. Returning a Genomic Result for an Adult-Onset Condition to the Parents of a Newborn: Insights From the BabySeq Project. Pediatrics. 2019 Jan;143(Suppl 1):S37-S43. doi: 10.1542/peds.2018-1099H. PMID 30600270
- [Background] VanNoy GE, Genetti CA, McGuire AL, Green RC, Beggs AH, Holm IA; BabySeq Project Group. Challenging the Current Recommendations for Carrier Testing in Children. Pediatrics. 2019 Jan;143(Suppl 1):S27-S32. doi: 10.1542/peds.2018-1099F. PMID 30600268
- [Background] Lu CY, Hendricks-Sturrup RM, Mazor KM, McGuire AL, Green RC, Rehm HL. The case for implementing sustainable routine, population-level genomic reanalysis. Genet Med. 2020 Apr;22(4):815-816. doi: 10.1038/s41436-019-0719-3. Epub 2019 Dec 12. No abstract available. PMID 31831882
- [Background] Mackay ZP, Dukhovny D, Phillips KA, Beggs AH, Green RC, Parad RB, Christensen KD; BabySeq Project Team. Quantifying Downstream Healthcare Utilization in Studies of Genomic Testing. Value Health. 2020 May;23(5):559-565. doi: 10.1016/j.jval.2020.01.017. Epub 2020 Mar 20. PMID 32389220
- [Derived] Armstrong B, Christensen KD, Genetti CA, Parad RB, Robinson JO, Blout Zawatsky CL, Zettler B, Beggs AH, Holm IA, Green RC, McGuire AL, Smith HS, Pereira S; BabySeq Project Team. Parental Attitudes Toward Standard Newborn Screening and Newborn Genomic Sequencing: Findings From the BabySeq Study. Front Genet. 2022 Apr 27;13:867371. doi: 10.3389/fgene.2022.867371. eCollection 2022. PMID 35571041
- [Derived] Pereira S, Smith HS, Frankel LA, Christensen KD, Islam R, Robinson JO, Genetti CA, Blout Zawatsky CL, Zettler B, Parad RB, Waisbren SE, Beggs AH, Green RC, Holm IA, McGuire AL; BabySeq Project Team. Psychosocial Effect of Newborn Genomic Sequencing on Families in the BabySeq Project: A Randomized Clinical Trial. JAMA Pediatr. 2021 Nov 1;175(11):1132-1141. doi: 10.1001/jamapediatrics.2021.2829. PMID 34424265
- [Derived] Schwartz TS, Christensen KD, Uveges MK, Waisbren SE, McGuire AL, Pereira S, Robinson JO, Beggs AH, Green RC; BabySeq Project Team; Bachmann GA, Rabson AB, Holm IA. Effects of participation in a U.S. trial of newborn genomic sequencing on parents at risk for depression. J Genet Couns. 2022 Feb;31(1):218-229. doi: 10.1002/jgc4.1475. Epub 2021 Jul 26. PMID 34309124
- [Derived] Knapp B, Decker C, Lantos JD. Neonatologists' Attitudes About Diagnostic Whole-Genome Sequencing in the NICU. Pediatrics. 2019 Jan;143(Suppl 1):S54-S57. doi: 10.1542/peds.2018-1099J. PMID 30600272
- See also: Related Info — https://www.genomes2people.org/research/babyseq/

RESULTS

PARTICIPANT FLOW:
Groups:
- Well Baby Parents: Family History Only: Parents of newborns in well-baby units receive an Annotated Family History Report only. Active Comparator: Standard of Care Only: Family History report only. Parents and their newborns are enrolled.
  Family history report: Participants from all arms of the study have a family history taken by a study genetic counselor. Information collected through the family history is summarized in a family history report tand reviewed with all participants.
- Well Babies: Family History Only: Newborns in well-baby units receive an Annotated Family History Report only. Active Comparator: Standard of Care Only: Family History report only. Parents and their newborns are enrolled.
  Family history report: Participants from all arms of the study have a family history taken by a study genetic counselor. Information collected through the family history is summarized in a family history report tand reviewed with all participants.
- Well Baby Parents: Family History + Exome Sequencing: Parents of newborns in well-baby units receive a Genome Report and an Annotated Family History Report. Main Study Experimental: Genome Report and Family History report. Parents and their newborns are enrolled.
  Genomic sequencing: Both sick and healthy infants randomized to receive genomic sequencing receive a 'Genomic Newborn Sequencing Report' (GNSR) which includes pathogenic or likely pathogenic variants identified in genes associated with childhood-onset disease.
  Family history report: Participants from all arms of the study have a family history taken by a study genetic counselor. Information collected through the family history is summarized in a family history report that is reviewed with all participants.
- Well Babies: Family History + Exome Sequencing: Newborns in well-baby units receive a Genome Report and an Annotated Family History Report. Main Study Experimental: Genome Report and Family History report. Parents and their newborns are enrolled.
  Genomic sequencing: Both sick and healthy infants randomized to receive genomic sequencing receive a 'Genomic Newborn Sequencing Report' (GNSR) which includes pathogenic or likely pathogenic variants identified in genes associated with childhood-onset disease.
  Family history report: Participants from all arms of the study have a family history taken by a study genetic counselor. Information collected through the family history is summarized in a family history report that is reviewed with all participants.
- ICU Baby Parents: Family History Only: Parents of newborns in intensive care units receive an Annotated Family History Report only. Active Comparator: Standard of Care Only: Family History report only. Parents and their newborns are enrolled.
  Family history report: Participants from all arms of the study have a family history taken by a study genetic counselor. Information collected through the family history is summarized in a family history report that is reviewed with all participants.
- ICU Babies: Family History Only: Newborns in intensive care units receive an Annotated Family History Report only. Active Comparator: Standard of Care Only: Family History report only. Parents and their newborns are enrolled.
  Family history report: Participants from all arms of the study have a family history taken by a study genetic counselor. Information collected through the family history is summarized in a family history report that is reviewed with all participants.
- ICU Baby Parents: Family History + Exome Sequencing: Parents of newborns in intensive care units receive a Genome Report and an Annotated Family History Report. Main Study Experimental: Genome Report and Family History report. Parents and their newborns are enrolled.
  Genomic sequencing: Both sick and healthy infants randomized to receive genomic sequencing receive a 'Genomic Newborn Sequencing Report' (GNSR) which includes pathogenic or likely pathogenic variants identified in genes associated with childhood-onset disease.
  Family history report: Participants from all arms of the study have a family history taken by a study genetic counselor. Information collected through the family history is summarized in a family history report that is reviewed with all participants.
- ICU Babies: Family History + Exome Sequencing: Newborns in intensive care units receive a Genome Report and an Annotated Family History Report. Main Study Experimental: Genome Report and Family History report. Parents and their newborns are enrolled.
  Genomic sequencing: Both sick and healthy infants randomized to receive genomic sequencing receive a 'Genomic Newborn Sequencing Report' (GNSR) which includes pathogenic or likely pathogenic variants identified in genes associated with childhood-onset disease.
  Family history report: Participants from all arms of the study have a family history taken by a study genetic counselor. Information collected through the family history is summarized in a family history report that is reviewed with all participants.
Period: Overall Study
Arm/Group | Well Baby Parents: Family History Only | Well Babies: Family History Only | Well Baby Parents: Family History + Exome Sequencing | Well Babies: Family History + Exome Sequencing | ICU Baby Parents: Family History Only | ICU Babies: Family History Only | ICU Baby Parents: Family History + Exome Sequencing | ICU Babies: Family History + Exome Sequencing
Started (Start is the number of participants (including parents and their newborns) who were randomized. Parents were enrolled with their newborns and at least one parent had to complete a baseline survey to be randomized into the study and considered fully enrolled.) | 255 | 128 | 257 | 129 | 66 | 33 | 68 | 34
Received Disclosure (Parents received disclosure for their newborns study results and responded to a post-disclosure survey. Either parent could complete or skip the survey.) | 158 | 79 (Newborns did not receive disclosure) | 194 | 97 | 43 | 21 | 38 | 19
Completed (Parents completed 10-month survey for their newborns. Either parent could complete or skip the survey.) | 143 | 0 (Newborns did not complete survey) | 168 | 0 (Newborns did not complete survey) | 39 | 0 (Newborns did not complete survey) | 38 | 0 (Newborns did not complete survey)
Not Completed | 112 | 128 | 89 | 129 | 27 | 33 | 30 | 34

BASELINE CHARACTERISTICS:
Groups:
- Well Baby Parents: Family History Only: Parents of newborns in well-baby units receive an Annotated Family History Report only. Active Comparator: Standard of Care Only: Family History report only
  Family history report: Participants from all arms of the study will have a family history taken by a study genetic counselor. Information collected through the family history will be summarized in a family history report that will be reviewed with all participants.
- Well Babies: Family History Only: Newborns in well-baby units receive an Annotated Family History Report only. Active Comparator: Standard of Care Only: Family History report only
  Family history report: Participants from all arms of the study will have a family history taken by a study genetic counselor. Information collected through the family history will be summarized in a family history report that will be reviewed with all participants.
- Well Baby Parents: Family History + Exome Sequencing: Parents of newborns in well-baby units receive a Genome Report and an Annotated Family History Report. Main Study Experimental: Genome Report and Family History report
  Genomic sequencing: Both sick and healthy infants randomized to receive genomic sequencing will receive a 'Genomic Newborn Sequencing Report' (GNSR) which will include pathogenic or likely pathogenic variants identified in genes associated with childhood-onset disease.
  Family history report: Participants from all arms of the study will have a family history taken by a study genetic counselor. Information collected through the family history will be summarized in a family history report that will be reviewed with all participants.
- Well Babies: Family History + Exome Sequencing: Newborns in well-baby units receive a Genome Report and an Annotated Family History Report. Main Study Experimental: Genome Report and Family History report
  Genomic sequencing: Both sick and healthy infants randomized to receive genomic sequencing will receive a 'Genomic Newborn Sequencing Report' (GNSR) which will include pathogenic or likely pathogenic variants identified in genes associated with childhood-onset disease.
  Family history report: Participants from all arms of the study will have a family history taken by a study genetic counselor. Information collected through the family history will be summarized in a family history report that will be reviewed with all participants.
- ICU Baby Parents: Family History Only: Parents of newborns in intensive care units receive an Annotated Family History Report only. Active Comparator: Standard of Care Only: Family History report only
  Family history report: Participants from all arms of the study will have a family history taken by a study genetic counselor. Information collected through the family history will be summarized in a family history report that will be reviewed with all participants.
- ICU Babies: Family History Only: Newborns in intensive care units receive an Annotated Family History Report only. Active Comparator: Standard of Care Only: Family History report only
  Family history report: Participants from all arms of the study will have a family history taken by a study genetic counselor. Information collected through the family history will be summarized in a family history report that will be reviewed with all participants.
- ICU Baby Parents: Family History + Exome Sequencing: Parents of newborns in intensive care units receive a Genome Report and an Annotated Family History Report. Main Study Experimental: Genome Report and Family History report
  Genomic sequencing: Both sick and healthy infants randomized to receive genomic sequencing will receive a 'Genomic Newborn Sequencing Report' (GNSR) which will include pathogenic or likely pathogenic variants identified in genes associated with childhood-onset disease.
  Family history report: Participants from all arms of the study will have a family history taken by a study genetic counselor. Information collected through the family history will be summarized in a family history report that will be reviewed with all participants.
- ICU Babies: Family History + Exome Sequencing: Newborns in intensive care units receive a Genome Report and an Annotated Family History Report. Main Study Experimental: Genome Report and Family History report
  Genomic sequencing: Both sick and healthy infants randomized to receive genomic sequencing will receive a 'Genomic Newborn Sequencing Report' (GNSR) which will include pathogenic or likely pathogenic variants identified in genes associated with childhood-onset disease.
  Family history report: Participants from all arms of the study will have a family history taken by a study genetic counselor. Information collected through the family history will be summarized in a family history report that will be reviewed with all participants.
- Total: Total of all reporting groups
Arm/Group | Well Baby Parents: Family History Only | Well Babies: Family History Only | Well Baby Parents: Family History + Exome Sequencing | Well Babies: Family History + Exome Sequencing | ICU Baby Parents: Family History Only | ICU Babies: Family History Only | ICU Baby Parents: Family History + Exome Sequencing | ICU Babies: Family History + Exome Sequencing | Total
Number analyzed (Participants) | 255 | 128 | 257 | 129 | 66 | 33 | 68 | 34 | 970
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 128 | 0 | 129 | 0 | 33 | 0 | 34 | 324
  Between 18 and 65 years | 255 | 0 | 257 | 0 | 66 | 0 | 68 | 0 | 646
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 34 (4.45) | .025 (.016) | 35 (4.60) | .027 (.017) | 32 (5.29) | .055 (.039) | 35 (5.38) | .060 (.031) | 34 (4.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 66 | 129 | 63 | 33 | 15 | 34 | 17 | 487
  Male | 125 | 62 | 128 | 66 | 33 | 18 | 34 | 17 | 483
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 15 | 9 | 9 | 7 | 5 | 1 | 1 | 67
  Not Hispanic or Latino | 196 | 88 | 212 | 107 | 55 | 25 | 64 | 30 | 777
  Unknown or Not Reported | 39 | 25 | 36 | 13 | 4 | 3 | 3 | 3 | 126
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Asian | 28 | 10 | 31 | 8 | 2 | 0 | 4 | 1 | 84
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
  Black or African American | 12 | 9 | 8 | 2 | 3 | 2 | 1 | 0 | 37
  White | 194 | 89 | 185 | 79 | 57 | 27 | 57 | 27 | 715
  More than one race | 5 | 12 | 9 | 24 | 0 | 2 | 0 | 3 | 55
  Unknown or Not Reported | 15 | 7 | 24 | 16 | 4 | 2 | 4 | 2 | 74
Region of Enrollment [Number; unit: participants]
  United States | 255 | 128 | 257 | 129 | 66 | 33 | 69 | 34 | 647

OUTCOME MEASURES:

1. Primary Outcome: Downstream Health Care Costs Attributable to BabySeq Project Disclosure: Days of Inpatient Care
Description: Days spent in inpatient care from disclosure of randomization status / genomic sequencing results through 10 months post-disclosure. Services were identified through a combination of chart note review, medical record review and participant surveys.
Time Frame: From disclosure through 10 Months post-disclosure (approx. 15 months after baseline).
Population: The analysis population included infants enrolled in the BabySeq project. Data was not available for all participants due to withdrawal or non-responsiveness to follow up surveys.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Well Baby Family History Only: Newborns in well-baby units receive an Annotated Family History Report only. Active Comparator: Standard of Care Only: Family History report only
  Family history report: Participants from all arms of the study will have a family history taken by a study genetic counselor. Information collected through the family history will be summarized in a family history report that will be reviewed with all participants.
- Well Baby Family History + Exome Sequencing: Newborns in well-baby units receive a Genome Report and an Annotated Family History Report. Main Study Experimental: Genome Report and Family History report
  Genomic sequencing: Both sick and healthy infants randomized to receive genomic sequencing will receive a 'Genomic Newborn Sequencing Report' (GNSR) which will include pathogenic or likely pathogenic variants identified in genes associated with childhood-onset disease.
  Family history report: Participants from all arms of the study will have a family history taken by a study genetic counselor. Information collected through the family history will be summarized in a family history report that will be reviewed with all participants.
- ICU Baby Family History Only: Newborns in intensive care units receive an Annotated Family History Report only. Active Comparator: Standard of Care Only: Family History report only
  Family history report: Participants from all arms of the study will have a family history taken by a study genetic counselor. Information collected through the family history will be summarized in a family history report that will be reviewed with all participants.
- ICU Baby Family History + Exome Sequencing: Newborns in intensive care units receive a Genome Report and an Annotated Family History Report. Main Study Experimental: Genome Report and Family History report
  Genomic sequencing: Both sick and healthy infants randomized to receive genomic sequencing will receive a 'Genomic Newborn Sequencing Report' (GNSR) which will include pathogenic or likely pathogenic variants identified in genes associated with childhood-onset disease.
  Family history report: Participants from all arms of the study will have a family history taken by a study genetic counselor. Information collected through the family history will be summarized in a family history report that will be reviewed with all participants.
Arm/Group | Well Baby Family History Only | Well Baby Family History + Exome Sequencing | ICU Baby Family History Only | ICU Baby Family History + Exome Sequencing
Number analyzed (Participants) | 116 | 121 | 31 | 30
Days | 0.1 (0.4) | 0.0 (0.3) | 3.1 (12.9) | 3.8 (12.9)

2. Primary Outcome: Parents' Distress
Description: Parents' Distress was assessed using validated scales measuring Anxiety and Depression, and a novel item assessing Blame with responses ranging from 1 to 5. Higher scores indicate more distress. Anxiety per the Edinburgh Postnatal Depression Scale anxiety subscale (baseline, post-disclosure, and 3 months; scores ranging from 0 to 9); Anxiety per the Generalized Anxiety Disorder Scale-7 (3 months and 10 months; scores ranging from 0 to 21); Depression per the Edinburgh Postnatal Depression Scale (baseline, post-disclosure, and 3 months; scores ranging from 0 to 30); Depression per the Patient Health Questionnaire-9 (3 months and 10 months; scores ranging from 0 to 30); Self-blame per a novel item (3 months and 10 months)
Time Frame: From baseline through 10 post-disclosure, with time points varying by measure. (Post-disclosure approx. 5 months after baseline; 3-months approx. 8 months after baseline; 10-months approx. 15 months after baseline)
Population: The analysis population included parents of infants enrolled in the BabySeq project. Data was not available for all participants due to withdrawal or non-responsiveness to follow up surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Well Baby Family History Only | Well Baby Family History + Exome Sequencing | ICU Baby Family History Only | ICU Baby Family History + Exome Sequencing
Number analyzed (Participants) | 202 | 203 | 53 | 60
score on a scale
  Anxiety per the Edinburgh Postnatal Depression Scale anxiety subscale - baseline | 2.6 (1.83) | 2.75 (1.83) | 3.04 (2.1) | 3.28 (2.05)
  Anxiety per the Edinburgh Postnatal Depression Scale anxiety subscale - Postdisclosure | 2.19 (1.86) | 2.34 (1.91) | 2.44 (2.29) | 2.56 (1.83)
  Anxiety per the Edinburgh Postnatal Depression Scale anxiety subscale - 3 months | 1.86 (1.87) | 1.97 (1.86) | 2.16 (2.07) | 2.24 (1.83)
  Anxiety per the Generalized Anxiety Disorder Scale-7 - 3 months | 2.4 (2.99) | 2.47 (2.83) | 3.34 (3.77) | 3.72 (4.52)
  Anxiety per the Generalized Anxiety Disorder Scale-7 - 10 months | 2.46 (3.06) | 2.77 (3.10) | 3.43 (4.2) | 2.25 (2.92)
  Depression per the Edinburgh Postnatal Depression Scale - baseline | 4.68 (3.62) | 4.96 (3.64) | 6.51 (4.69) | 6.69 (4.72)
  Depression per the Edinburgh Postnatal Depression Scale - postdisclosure | 4.12 (3.51) | 4.38 (3.85) | 5.0 (5.03) | 4.92 (4.54)
  Depression per the Edinburgh Postnatal Depression Scale - 3 months | 3.53 (3.45) | 3.96 (3.68) | 5.13 (4.90) | 4.54 (4.33)
  Depression per the Patient Health Questionnaire-9 - 3 months | 4.04 (3.47) | 3.49 (2.79) | 4.86 (5.93) | 4.35 (3.20)
  Depression per the Patient Health Questionnaire-9 - 10 months | 3.79 (3.04) | 3.96 (3.21) | 5.20 (6.25) | 4.42 (3.05)
  novel item assessing Blame - 3 months | 1.8 (0.83) | 1.96 (0.90) | 2.12 (0.93) | 1.97 (0.811)
  novel item assessing Blame - 10 months | 1.95 (0.89) | 1.78 (0.86) | 2.39 (1.10) | 1.87 (0.70)

3. Primary Outcome: Parent-Child Relationship
Description: Parent-Child Relationship was assessed using validated scales measuring parents' perceptions of parenting stress (General parenting stress per the Parenting Stress Index™, 4th Edition Short Form (10 months); scores range from 36 to 180), how vulnerable they perceive their child to be (Parents' perception of baby's vulnerability per the Vulnerable Baby Scale (baseline, postdisclosure, 3 months, 10 months); scores range from 4 to 20), and how they are bonding with their child (Parent-child bonding per the Mother-to-Infant Bonding Scale (baseline, postdisclosure, 3 months, 10 months); scores range from 0 to 24). Lower bonding scores indicate more problems with bonding. For other measures, higher scores indicate higher stress and perceptions of vulnerability.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Well Baby Family History Only | Well Baby Family History + Exome Sequencing | ICU Baby Family History Only | ICU Baby Family History + Exome Sequencing
Number analyzed (Participants) | 212 | 212 | 54 | 63
score on a scale
  Parent-child bonding per the Mother-to-Infant Bonding Scale - baseline | 1.6 (1.83) | 1.35 (1.82) | 1.45 (1.76) | 1.71 (1.65)
  Parent-child bonding per the Mother-to-Infant Bonding Scale - postdisclosure | 1.18 (1.64) | 1.15 (1.45) | 1.05 (1.25) | 0.95 (1.21)
  Parent-child bonding per the Mother-to-Infant Bonding Scale - 3 months | 1.48 (1.79) | 1.36 (1.63) | 1.56 (1.90) | 1.03 (1.36)
  Parent-child bonding per the Mother-to-Infant Bonding Scale - 10 months | 1.47 (1.81) | 1.45 (1.81) | 1.74 (3.14) | 1.30 (1.57)
  Vulnerable Baby Scale - baseline | 9.02 (2.82) | 9.11 (2.82) | 13.01 (3.88) | 13.54 (3.58)
  Vulnerable Baby Scale - postdisclosure | 8.03 (2.44) | 8.59 (2.79) | 10.24 (3.37) | 11.55 (3.72)
  Vulnerable Baby Scale - 3 months | 8.17 (2.63) | 8.27 (2.79) | 9.77 (3.61) | 9.84 (3.32)
  Vulnerable Baby Scale - 10 months | 7.3 (2.3) | 7.46 (2.32) | 8.51 (3.06) | 9.21 (3.14)
  Parenting Stress Index™, 4th Edition Short Form- 10 months | 61.17 (18.19) | 60.46 (15.55) | 64.94 (19.15) | 62.03 (15.11)

4. Primary Outcome: Parents' Relationship
Description: Parents' Relationship was assessed using validated and novel measures of marital satisfaction using the Relationship satisfaction per the Kansas Marital Satisfaction Scale (3 months; scores ranging from 3 to 15), relationship conflict per a novel item (all time points; scores ranging from 1 to 5), and partner blame per a novel item (3 months and 10 months; scores ranging from 1 to 5). Higher scores on Satisfaction indicates more Satisfaction. Higher scores on Conflict and Blame indicate higher conflict and blame.
Time Frame: From baseline through 10 post-disclosure, with time points varying by measure. Post-disclosure approx. 5 months after baseline; 3-months approx. 8 months after baseline; 10-months approx. 15 months after baseline.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Well Baby Family History Only | Well Baby Family History + Exome Sequencing | ICU Baby Family History Only | ICU Baby Family History + Exome Sequencing
Number analyzed (Participants) | 210 | 210 | 55 | 62
score on a scale
  Kansas Marital Satisfaction Scale - 3 months | 15.0 (2.47) | 13.14 (2.12) | 12.94 (2.12) | 12.92 (2.34)
  relationship conflict - baseline | 1.92 (0.77) | 1.99 (0.75) | 2.01 (0.80) | 1.87 (0.76)
  relationship conflict - postdisclosure | 2.01 (0.74) | 2.09 (0.75) | 1.89 (0.77) | 2.02 (0.76)
  relationship conflict - 3 months | 2.0 (0.74) | 2.17 (0.74) | 2.05 (0.90) | 2.02 (0.75)
  relationship conflict - 10 months | 2.09 (0.83) | 2.21 (0.78) | 2.27 (1.12) | 2.04 (0.82)
  partner blame 3 months | 1.69 (0.64) | 1.86 (0.81) | 2.03 (0.85) | 1.85 (0.71)
  partner blame 10 months | 1.87 (0.79) | 1.72 (0.71) | 2.13 (0.91) | 1.71 (0.46)

5. Primary Outcome: Downstream Health Care Utilization Attributable to BabySeq Project Disclosure: Number of Health Care Provider Visits
Description: Per-patient counts for number of health care provider visits. Services were identified through a combination of chart note review, medical record review and participant surveys.
Time Frame: From disclosure through 10 Months post-disclosure (approx. 15 months after baseline)
Measure: Mean (Standard Deviation); unit: # of Visits
Arm/Group | Well Baby Family History Only | Well Baby Family History + Exome Sequencing | ICU Baby Family History Only | ICU Baby Family History + Exome Sequencing
Number analyzed (Participants) | 116 | 121 | 31 | 30
# of Visits | 5.4 (6.3) | 5.9 (6.1) | 4.9 (7.4) | 6.3 (7.2)

6. Primary Outcome: Downstream Health Care Utilization Attributable to BabySeq Project Disclosure: Number of Current Medications at 10 Months
Description: Per-patient counts for number of current medications at 10 months. Services were identified through a combination of chart note review, medical record review and participant surveys.
Time Frame: From disclosure through 10 Months post-disclosure (approx. 15 months after baseline)
Measure: Mean (Standard Deviation); unit: # of current medications at 10 mont
Arm/Group | Well Baby Family History Only | Well Baby Family History + Exome Sequencing | ICU Baby Family History Only | ICU Baby Family History + Exome Sequencing
Number analyzed (Participants) | 116 | 121 | 31 | 30
# of current medications at 10 mont | 1.7 (4.9) | 1.4 (3.2) | 0.5 (1.0) | 1.8 (4.0)

7. Primary Outcome: Downstream Health Care Utilization Attributable to BabySeq Project Disclosure: Number of ER Visits
Description: Per-patient counts number of ER visits. Services were identified through a combination of chart note review, medical record review and participant surveys.
Time Frame: From disclosure through 10 Months post-disclosure (approx. 15 months after baseline)
Measure: Mean (Standard Deviation); unit: # of ER visits
Arm/Group | Well Baby Family History Only | Well Baby Family History + Exome Sequencing | ICU Baby Family History Only | ICU Baby Family History + Exome Sequencing
Number analyzed (Participants) | 116 | 121 | 31 | 30
# of ER visits | 0.3 (0.7) | 0.4 (0.8) | 0.5 (1.1) | 0.3 (0.7)

8. Primary Outcome: Downstream Health Care Utilization Attributable to BabySeq Project Disclosure: Number of Outpatient Lab Tests
Description: Per-patient counts for number of outpatient lab tests after results disclosure. Services were identified through a combination of chart note review, medical record review and participant surveys.
Time Frame: From disclosure through 10 Months post-disclosure (approx. 15 months after baseline)
Measure: Mean (Standard Deviation); unit: # of Outpatient Lab Tests
Arm/Group | Well Baby Family History Only | Well Baby Family History + Exome Sequencing | ICU Baby Family History Only | ICU Baby Family History + Exome Sequencing
Number analyzed (Participants) | 116 | 121 | 31 | 30
# of Outpatient Lab Tests | 0.2 (1.1) | 0.1 (0.6) | 0.0 (0.2) | 0.1 (0.4)

9. Primary Outcome: Downstream Health Care Utilization Attributable to BabySeq Project Disclosure
Description: Per-patient means (SDs) for healthcare costs (in U.S. dollars) after disclosure of randomization status / genomic results from the BabySeq project. Services were identified through a combination of chart note review, medical record review and participant surveys.
Time Frame: From disclosure through 10 Months post-disclosure (approx. 15 months after baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U.S. dollars
Arm/Group | Well Baby Family History Only | Well Baby Family History + Exome Sequencing | ICU Baby Family History Only | ICU Baby Family History + Exome Sequencing
Number analyzed (Participants) | 116 | 121 | 31 | 30
U.S. dollars
  Cost of Days Inpatient / Inpatient Care | 424 (2230) | 301 (2389) | 23472 (114624) | 25012 (87820)
  Cost of Visits / Outpatient services | 1348 (1645) | 1440 (1623) | 1144 (1603) | 1762 (2261)
  Cost of Med # / Medications (OOP) | 24 (85) | 17 (57) | 1194 (6587) | 45 (95)
  Cost of ER Visits / Equipment (OOP) | 176 (312) | 200 (400) | 62 (105) | 72 (158)
  Cost of Labs / Total | 1972 (3305) | 1958 (3019) | 25872 (114756) | 26891 (87456)

10. Secondary Outcome: Change in Perceived Utility Toward Genomic Sequencing
Description: A novel survey item asked participants to rate the usefulness of whole genome sequencing results for managing health on a 1-10 scale at baseline and 3 months post-disclosure. Responses were on a 10-point scale anchored by "not at all useful" (1) to "extremely useful" (10).
Time Frame: From Baseline to 3 Months post-disclosure (approx. 8 months after baseline)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Well Baby Family History Only | Well Baby Family History + Exome Sequencing | ICU Baby Family History Only | ICU Baby Family History + Exome Sequencing
Number analyzed (Participants) | 201 | 204 | 53 | 60
score on a scale
  perceived utility - baseline | 3.78 (0.86) | 3.77 (0.95) | 4.13 (0.81) | 3.76 (1.02)
  perceived utility - 3 months | 3.83 (0.91) | 4.23 (0.83) | 4.10 (0.79) | 4.25 (0.77)

11. Other Pre Specified Outcome: Understanding
Description: A novel item assessed participants' subjective understanding of their study results on a 1-5 scale, where higher scores indicate greater subjective understanding.
Time Frame: Post-disclosure approx. 5 months after baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Well Baby Family History Only | Well Baby Family History + Exome Sequencing | ICU Baby Family History Only | ICU Baby Family History + Exome Sequencing
Number analyzed (Participants) | 143 | 163 | 35 | 35
score on a scale | 3.69 (0.55) | 3.37 (0.70) | 3.51 (0.70) | 3.14 (0.60)

ADVERSE EVENTS:
Time Frame: From enrollment through 10 months after disclosure of family history and/or newborn genomic sequencing results to families.
Description: Any serious adverse events linked to the disclosure of genomic information will be reported both to the Institutional Review Board (IRB) and the Data Safety Monitoring Board (DSMB) at the time the event is identified. For all other metrics, the DSMB will review data annually: statistics, decline and drop-out rates and reasons, as well as any non-serious adverse events (e.g. changes in anxiety or distress scales that do not rise to the level of serious adverse events).
Arm/Group | Well Baby Parents: Family History Only | Well Babies: Family History Only | Well Baby Parents: Family History + Exome Sequencing | Well Babies: Family History + Exome Sequencing | ICU Baby Parents: Family History Only | ICU Babies: Family History Only | ICU Baby Parents: Family History + Exome Sequencing | ICU Babies: Family History + Exome Sequencing
All-Cause Mortality (participants affected / at risk) | 0/255 | 0/128 | 0/257 | 0/129 | 0/66 | 0/33 | 0/68 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/255 | 0/128 | 0/257 | 0/129 | 0/66 | 0/33 | 0/68 | 0/34
Other Adverse Events (participants affected / at risk) | 0/255 | 0/128 | 0/257 | 0/129 | 0/66 | 0/33 | 0/68 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/11/NCT02422511/Prot_SAP_000.pdf